CLINICAL TRIAL: NCT00815139
Title: Evaluation in 3 moNths Duration of nEointimAl coVerAge After zOtaRolimus-Eluting Stent Implantation by Optical Coherence Tomography (ENDEAVOR OCT)
Brief Title: Evaluation of Zotarolimus Eluting Stent at 3 Months Using Optical Coherence Tomography
Acronym: ENDEAVOR OCT
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Yangsoo Jang, Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei Univerisity
Other Study IDs: 4-2007-0409
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease, stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ZES group: Groups who were treated with zotarolimus eluting stent

SUMMARY:
Neointimal coverage over stent strut is important for preventing the stent thrombosis. But, there is no data for the duration of complete formation of neointima om zotarolimus eluting stent (ZES). Previously the investigational observational data at 9 months showed most of stent strut was covered with neointima. Therefore, the investigators investigated the evaluation of neointimal coverage on 3 months after ZES implantation using novel OCT system, which is powerful intravascular imaging system having the higher resolution power.

DETAILED DESCRIPTION:
Stent thrombosis is current main issue after introduction of drug-eluting stents and theoretically dual antiplatelet therapy should be continued to prevent the stent thrombosis until complete reendothelization. Currently, AHA/ACC guideline recommend dual antiplatelet should continue at least 3 months in Sirolimus eluting stent (SES) and 6 months in paclitaxel eluting stent (PES), but if possible, suggest to use until 12 months.

Zotarolimus (Endeavor®) eluting stent (ZES) have been recently introduced and focused on reducing concern of safety through the biocompatible polymer and rapid drug elution. ENDEAVOR II trial showed a 0.5 per cent rate of stent thrombosis at 30 days - with no late thrombosis beyond 30 days and no late stent malapposition. In the long term follow up data of Endeavor stent, the two-year clinical results of ENDEAVOR I were impressive, with a low TVF and MACE rate (2% and 3% respectively) with the absence of reported thromboses after day 14. These results speak, especially the lack of stent thrombosis after 14 days, reflect very well on the performance and safety of the ZES.

But, there has been no guideline for the duration of dual antiplatelet therapy in ZES although shorter duration of dual antiplatelet therapy could be safe compared to previous drug-eluting stents. Also, there is no data how long duration might be taken in completion of reendothelialization after ZES implantation in living patients. The most powerful histological predictor of stent thrombosis was endothelial coverage. The best morphometric predictor of LST was the ratio of uncovered to total stent struts. Because the presence of endothelization is not available in in vivo situation and endothelialization is reported to be associated with neointimal coverage of stent, the detection of neointima after stent implantation could be the main issue to predict the stent thrombosis. Recent data in SES using optical coherence tomography (OCT) reported neointimal coverage over a SES at 3-month follow-up is incomplete. The rates of exposed struts and exposed struts with malapposition were 15% and 6%, respectively. These were more frequent in patients with acute coronary syndrome (ACS) than in those with non-ACS (18% vs 13%, p <0.0001; 8% vs 5%, p <0.005, respectively).

Although neointimal coverage could be completely in early period after ZES implantation, there is no data for this finding. Therefore, we investigate the evaluation of neointimal coverage on 3 months after ZES implantation using novel OCT system, which is powerful intravascular imaging system having the higher resolution power. This study may provide adequate information on the safety of discontinuation of dual antiplatelet therapy for patients in clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Significant coronary de novo lesion ( > 70% by quantitative angiographic analysis)
* Patients with stable or acute coronary syndrome considered for coronary revascularization.
* Non-emergent conditions
* Reference vessel diameter of 2.75 to 4.0 mm by operator assessment

Exclusion Criteria:

* The criteria for exclusion were contraindication to anti-platelet agents
* ST elevation MI requiring primary PCI
* Proximal lesion within 15 mm from ostium
* Prior insertion of other DES in any vessel
* Creatinine level more than 2.0mg/dL or ESRD
* Severe hepatic dysfunction (more than 3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy less than 1 year
* Complex lesion morphologies (aorto-ostial, bifurcation with >2.0 mm side branch, unprotected Left main, thrombus, severe calcification, chronic total occlusion)
* Target lesion is vein graft lesion
* Reference vessel <2.5 mm or >4.0 mm diameter by visual estimation
* Long lesion that require more than two stents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the cath lab for non-emergent percutaenous coronary intervention and stenting are eligible for participation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to evaluate the neointimal coverage of Zotarolimus (Endeavor®) eluting stent (ZES) in 3 month after stent implantation by Optical coherence tomography. | 3 months

SECONDARY OUTCOMES:
to compare the difference in neointimal coverage between ACS and non-ACS and to compare the difference in detection of neointimal coverage between OCT and IVUS at 3 months. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yangsoo Jang, MD, Ph D, Principal Investigator — Division of Cardiology, Cardiovascular Hospital, Yonsei University
Locations (1):
- Division of Cardiology, Cardiovascular Hospital, Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Kim JS, Jang IK, Fan C, Kim TH, Kim JS, Park SM, Choi EY, Lee SH, Ko YG, Choi D, Hong MK, Jang Y. Evaluation in 3 months duration of neointimal coverage after zotarolimus-eluting stent implantation by optical coherence tomography: the ENDEAVOR OCT trial. JACC Cardiovasc Interv. 2009 Dec;2(12):1240-7. doi: 10.1016/j.jcin.2009.10.006. PMID 20129551